CLINICAL TRIAL: NCT02916225
Title: High Intensity Interval Training Versus Moderate Continuous Training in Heart Failure With Preserved Ejection Fraction Patients: a Randomized Study.
Brief Title: High Intensity Interval Training Versus Moderate Continuous Training in Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Ricardo Stein, Assistant Professor, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140362
Record Dates: First submitted 2016-09-25; First posted 2016-09-27 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure; Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity interval training (Active Comparator): exercise protocol for high intensity/aerobic interval training as described by ESC statement (Mezzani et al.)
  Interventions: Behavioral: High Intensity Interval Training
- Moderate Continuous Training (Placebo Comparator): exercise protocol for continuous aerobic training as described by ESC statement (Mezzani et al.)
  Interventions: Behavioral: Moderate Continuous Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — The HIIT group will warm up for 10 minutes at 60% to 70% of peak heart rate(50% to 60% of V̇O2peak) before walking four 4-minute intervals at 85% to 95% of peak heart rate. Each interval will be separated by 3-minute active pauses, walking at 60% to 70% of peak heart rate. The training session will be terminated by a 3-minute cool-down at 60% to 70% of peak heart rate. Total exercise time will be 38 minutes for the HIIT group. Patients will perform 3 training sessions per week for 12 consecutive weeks.
  Arms: High intensity interval training
Behavioral: Moderate Continuous Training — The moderate continuous training (MCT) group will undergo treadmill walking continuously at 60% to 70% of peak heart rate for 47 minutes each session to make sure the training protocols will be isocaloric. Patients will perform 3 training sessions per week for 12 consecutive weeks.
  Arms: Moderate Continuous Training

SUMMARY:
The purpose of this study is to determine whether high intensity interval training (HIIT) is superior to moderate continuous training in increasing cardiopulmonary capacity in heart failure with preserved ejection fraction patients.

DETAILED DESCRIPTION:
High intensity interval training (HIIT) has been proved to increase oxygen consumption, having superior cardiovascular effect when compared to moderate continuous training (MCT) in post-infarction patients (Wisloff et al.) Aerobic training also had shown positive effect on oxygen consumption and diastolic function in subjects with HFPEF when compared to usual care (Edelmann et al).

However, the comparison of HIIT and MCT on improving functional capacity and diastolic function in HFPEF patients has not yet been study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure with preserved ejection fraction (HFPEF) of any etiology that have functional class of the New York Heart Association (NYHA) between I and III, left ventricular ejection fraction > 50% and who meet clinical and echocardiography criteria for HFPEF according to the consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology (Paulus et al.). Patients should be clinical stable for the last 3 months and under optimized pharmacologic treatment, being capable of walking without limitations.

Exclusion Criteria:

* Patients with exercise-induced unstable ventricular arrhythmias, unstable angina, moderate to severe valvular heart disease, severe pulmonary disease, severe anemia, cognitive limitations to understand study protocol, use of pacemaker, autonomic neuropathy, cardiovascular event for less than 3 months, congenital heart disease, terminal illness with less than 1 year of life expectancy, peripheral arterial disease with intermittent claudication or osteoarticular conditions limiting exercise will be excluded.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Consumption | 12 weeks after beginning of training

SECONDARY OUTCOMES:
Diastolic Function | 12 weeks after beginning of training
  assessed by echocardiography
Pulmonary function tests | 12 weeks after beginning of training
  assessed by spirometry
Respiratory muscle strength | 12 weeks after beginning of training
  assessed by manovacuometry
Quality of life | 12 weeks after beginning of training
  Minnesota Living with Heart Failure Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, ScD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mezzani A, Hamm LF, Jones AM, McBride PE, Moholdt T, Stone JA, Urhausen A, Williams MA; European Association for Cardiovascular Prevention and Rehabilitation; American Association of Cardiovascular and Pulmonary Rehabilitation; Canadian Association of Cardiac Rehabilitation. Aerobic exercise intensity assessment and prescription in cardiac rehabilitation: a joint position statement of the European Association for Cardiovascular Prevention and Rehabilitation, the American Association of Cardiovascular and Pulmonary Rehabilitation and the Canadian Association of Cardiac Rehabilitation. Eur J Prev Cardiol. 2013 Jun;20(3):442-67. doi: 10.1177/2047487312460484. Epub 2012 Oct 26. PMID 23104970
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822
- [Background] Edelmann F, Gelbrich G, Dungen HD, Frohling S, Wachter R, Stahrenberg R, Binder L, Topper A, Lashki DJ, Schwarz S, Herrmann-Lingen C, Loffler M, Hasenfuss G, Halle M, Pieske B. Exercise training improves exercise capacity and diastolic function in patients with heart failure with preserved ejection fraction: results of the Ex-DHF (Exercise training in Diastolic Heart Failure) pilot study. J Am Coll Cardiol. 2011 Oct 18;58(17):1780-91. doi: 10.1016/j.jacc.2011.06.054. PMID 21996391
- [Derived] Donelli da Silveira A, Beust de Lima J, da Silva Piardi D, Dos Santos Macedo D, Zanini M, Nery R, Laukkanen JA, Stein R. High-intensity interval training is effective and superior to moderate continuous training in patients with heart failure with preserved ejection fraction: A randomized clinical trial. Eur J Prev Cardiol. 2020 Nov;27(16):1733-1743. doi: 10.1177/2047487319901206. Epub 2020 Jan 21. PMID 31964186